CLINICAL TRIAL: NCT05857202
Title: Oxidative Stress and Inflammation Biomarkers in Correlation to Postoperative Pain Modulation in Surgically Treated Patients With Laryngeal Cancer
Brief Title: Oxidative Stress and Inflammation Biomarkers in Surgically Treated Patients With Laryngeal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinical Centre of Serbia (Other)
Collaborators: University of Belgrade (Other)
Responsible Party: Principal Investigator, Ana Jotić, Assistant professor, MD, PhD, Clinical Centre of Serbia
Other Study IDs: 754/5
Record Dates: First submitted 2023-03-29; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Oxidative Stress Induction; Laryngeal Cancer; Interleukins; Pain Management; Quality of Life; Pain, Postoperative
Keywords: oxidative stress; laryngeal cancer; pain management; interleukins
MeSH Terms: conditions — Laryngeal Neoplasms; Agnosia; Pain, Postoperative | interventions — Analgesics, Opioid; Analgesics, Non-Narcotic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples that were taken from the patients for the analysis of oxidative stress (glutathione peroxidase 1, superoxide dismutase 1 and malondialdehyde) parameters and inflammation parameters (interleukin 1 and 6) before the operative treatment and after the operative treatment (1 postoperative day and 7 postoperative day).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Operated laryngeal cancer patients treated with non narcotic: Operated laryngeal cancer patients who were administered non narcotic drugs postoperative for pain management
  Interventions: Drug: Analgesics, Non-Narcotic
- Operated laryngeal cancer patients treated with non narcotic and opioids: Operated laryngeal cancer patients who were administered non narcotic and opioids postoperative for pain management
  Interventions: Drug: Analgesics, Opioid; Drug: Analgesics, Non-Narcotic
- Operated laryngeal cancer patients treated with opioids: Operated laryngeal cancer patients who were administered opioids postoperative for pain management
  Interventions: Drug: Analgesics, Opioid

INTERVENTIONS:
Drug: Analgesics, Opioid — Drugs were given immediately after the surgery, and correlation between analgesic use and parameters of oxidative stress and inflammation was assessed.
  Groups: Operated laryngeal cancer patients treated with non narcotic and opioids; Operated laryngeal cancer patients treated with opioids
Drug: Analgesics, Non-Narcotic — Drugs were given immediately after the surgery, and correlation between analgesic use and parameters of oxidative stress and inflammation was assessed.
  Groups: Operated laryngeal cancer patients treated with non narcotic; Operated laryngeal cancer patients treated with non narcotic and opioids

SUMMARY:
A experimental interventional prospective study will include patients with squamocellular carcinoma of the larynx surgically treated at the tertiary referral center. Clinical and demographic characteristics of the patients would be noted. The visual analog scale (VAS), Brief Pain Inventory questionnaire, Diagnosing Neuropathic Pain 4 (DN4) and Pain Detect Questionnaire were used for pain assessment. Questionnaire Quality of Life in Head and Neck Cancer Patients (QLQ - H&N35) was used to assess the quality of life in patients with surgically treated laryngeal carcinoma. The type and consumption of analgesics used after surgery was monitored. The analgesics were used according to WHO Ladder. Blood samples ware taken from the patients for the analysis of oxidative stress parameters and inflammation parameters before the operative treatment and after the operative treatment (1-2 postoperative day and 9-10 postoperative day). The concentrations of interleukin 1 (IL-1) and 6 (IL-6), glutathione peroxidase 1 (GPX1), superoxide dismutase 1 (SOD1) and malondialdehyde (MDA) in the serum were determined.

The aim of the study will be to assess concentrations of inflammatory biomarkers (IL-1, IL-6) and oxidative stress factors (MDA, SOD, GPKS1) in postoperative course in surgically treated patients with laryngeal carcinoma and in possible complication occurrence. Also, their correlation to type and dosage of used analgesics, to pain assessment questionnaire scores and QOL questionnaire scores in surgically treated patients with laryngeal carcinoma will be assessed.

DETAILED DESCRIPTION:
Patient selection

A experimental interventional prospective study would include 100 patients with squamocellular carcinoma of the larynx surgically treated in the period from October 2022 to February 2023 at the tertiary referral center. This study was approved by the Institutional Ethics Committee (745/5-22), and all patients signed the informed consent form prior to their inclusion in the study. The diagnosis of laryngeal carcinoma was confirmed by otorhinolaryngological clinical examination and laryngomicroscopic examination of the larynx with the biopsy and histopathologic examination of the tissue. Additional diagnostics (chest radiography and computed tomography of the neck and ultrasonography of the abdomen) were performed to determine the TNM stage of the disease. Study included patients with all stages of operable laryngeal carcinoma (T1-T4, N0-N2), without previous treated malignancies. Exclusion criteria were inoperable malignant disease, presence of distant metastases, previously treated malignancies, presence of neurological or other severe comorbidities which prevent surgical treatment, the presence of neurological or other severe physical and metabolic comorbidities, substance abuse, and the inability to provide informed consent.

The modality of treatment for every patient was decided on the institutional Oncological Board (consisting of a radiotherapist, head and neck surgeons, an oncologist, and a histopathologist). Open surgical treatment involved resection of the tumor (cordectomy, partial or total laryngectomy) with or without some form of the neck dissection in case of cervical lymphadenopathy. Demographic, clinical and histopathological characteristics (age and gender, tobacco use, histopathological tumor grade, TNM classification, and therapy modality) were noted.

Quality of life assessment

Questionnaire Quality of Life in Head and Neck Cancer Patients (QLQ - H&N35) was used to assess the quality of life in patients with surgically treated laryngeal carcinoma.

Pain assessment

The visual analog scale (VAS) was used for pain assessment. Scores were based on self-reported measures of pain severety that are recorded with a mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale (0 cm on the left end of the scale marks ''no pain'' and 10 cm on the right end of the scale marks ''the worst pain'').

Brief Pain Inventory questionnaire, Diagnosing Neuropathic Pain 4 (DN4) and Pain Detect Questionnaire were used for quality assessment of postoperative pain

Postoperative analgesia

The type and consumption of analgesics used after surgery was monitored. The analgesics were used according to WHO Ladder: (1) for mild to moderate pain, a non-opioid (acetaminophen or non-steroid anti-inflammatory drug , NSAID) with or without an adjuvant; (2) for moderate or severe pain, a non-opioid with an opioid for moderate pain and (3) an opioid for moderate to severe pain not combined with another agent.

Measurement of the Oxidative Stress and Inflammatory Parameters

Blood was taken from the patients for the analysis of oxidative stress parameters and inflammation parameters before the operative treatment and after the operative treatment (1-2 postoperative day and 9-10 postoperative day). The concentrations of interleukin 1 (IL-1) and 6 (IL-6), glutathione peroxidase 1 (GPX1), superoxide dismutase 1 (SOD1) and malondialdehyde (MDA) in the serum were determined by coated enzyme-linked immunosorbent assay (ELISA) kits, according to the manufacturer's instructions (Elabscience, Wuhan, China). The ELISA kits for determination of concentrations of IL-1 and IL-6 were based on the Sandwich ELISA principle, with plates pre-coated with an antibody specific to human cytokines. The optical density (OD) was measured spectrophotometrically at 450 nm, using a Multiskan EX plate reader (Thermo Fisher Scientific, Vantaa, Finland). The concentration of analytesin of the tested samples was calculated by comparing the OD of the samples to the standard curve created with GraphPad Prism 9.0 software (GraphPad Software Inc., San Diego, CA, USA).

Statistical analysis

Categorical data was described by absolute and relative numbers (in percentages), while numerical data was reported as arithmetic mean and standard deviation or median and interquartile range (IQR), depending on the data distribution. The normality was evaluated using mathematical (Shapiro-Willk, skewness and kurtosis, and coefficient of variation) and graphical (histogram, box plot) methods. For the evaluation of changing of pain intensity, parameters of oxidative stress, and biomarkers of inflammation Friedman test was applied with Wilcoxon signed rank test as post-hoc testing method. For analyzing the association between pain intensity (VAS), parameters of oxidative stress, and biomarkers of inflammation Spearman's rank correlation coefficient was used, because variables didn't have normal distribution. In order to evaluate all possible factors that influence the level of oxidative stress expressed as SOD and MDA levels, linear regression analysis (enter method) was performed reporting regression coefficient B, 95% confidence level (CI) of B, and p value. Univariate analysis was done first, and all significant factors were combined in multivariate models. All statistical methods were considered significant if p value was less or equal 0.05. The analysis was performed in IBM SPSS ver. 26.

ELIGIBILITY:
Inclusion Criteria:

* patients with all stages of diagnosed and operable laryngeal squamocellular carcinoma (T1-T4, N0-N2)

Exclusion Criteria:

* inoperable malignant disease
* presence of distant metastases
* previously treated malignancies
* presence of neurological or other severe comorbidities which prevent surgical treatment
* the presence of neurological or other severe physical and metabolic comorbidities
* substance abuse
* the inability to provide informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study would include 100 patients with squamocellular carcinoma of the larynx surgically treated at the tertiary referral center. The diagnosis of laryngeal carcinoma was confirmed by otorhinolaryngological clinical examination, laryngomicroscopic examination with the biopsy and histopathologic examination. Additional diagnostics (chest radiography and computed tomography of the neck and ultrasonography of the abdomen) were performed to determine the TNM stage of the disease.
  The modality of surgical treatment was decided on the institutional Oncological Board and involved resection of the tumor (cordectomy, partial or total laryngectomy) with or without some form of the neck dissection in case of cervical lymphadenopathy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between inflammatory marker IL-1 and pain intensity | 7 days
  A positive correlation between concentration of inflammatory marker IL-1 and pain intensity (VAS score) in postoperatively in surgically treated patients with laryngeal cancer is expected.
  The concentrations of inflammatory parameters IL-1 (pg/mL) in the blood serum were determined by ELISA kits, according to the manufacturer's instructions.
  Pain intensity would be assessed using the visual analog scale (VAS). Scores were based on self-reported measures of pain severity recorded with a mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale (0 mm on the left end of the scale marks ''no pain'' and 100mm on the right end of the scale marks ''the worst pain'').
  Correlation would be calculated with Spearman's rank correlation coefficient.
Correlation between inflammatory marker IL-6 and pain intensity | 7 days
  A positive correlation between concentration of inflammatory marker IL-6 and pain intensity (VAS score) in postoperatively in surgically treated patients with laryngeal cancer is expected.
  The concentrations of inflammatory marker IL-6 (pg/mL) in the blood serum were determined by ELISA kits, according to the manufacturer's instructions.
  Pain intensity would be assessed using the visual analog scale (VAS). Scores were based on self-reported measures of pain severity recorded with a mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale (0 mm on the left end of the scale marks ''no pain'' and 100mm on the right end of the scale marks ''the worst pain'').
  Correlation would be calculated with Spearman's rank correlation coefficient.
Correlation between inflammatory marker CRP and pain intensity | 7 days
  A positive correlation between concentration of inflammatory marker CRP and pain intensity (VAS score) in postoperatively in surgically treated patients with laryngeal cancer is expected.
  The concentrations of inflammatory marker CRP (ng/mL) in the blood serum were determined by ELISA kits, according to the manufacturer's instructions.
  Pain intensity would be assessed using the visual analog scale (VAS). Scores were based on self-reported measures of pain severity recorded with a mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale (0 mm on the left end of the scale marks ''no pain'' and 100mm on the right end of the scale marks ''the worst pain'').
  Correlation would be calculated with Spearman's rank correlation coefficient.
Correlation between oxidative stress marker MDA and pain intensity | 7 days
  A positive correlation between concentration of oxidative stress marker MDA and pain intensity (VAS score) in postoperatively in surgically treated patients with laryngeal cancer is expected.
  The concentrations of oxidative stress marker MDA (ng/mL) in the blood serum were determined by ELISA kits, according to the manufacturer's instructions.
  Pain intensity would be assessed using the visual analog scale (VAS). Scores were based on self-reported measures of pain severity recorded with a mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale (0 mm on the left end of the scale marks ''no pain'' and 100mm on the right end of the scale marks ''the worst pain'').
  Correlation would be calculated with Spearman's rank correlation coefficient.
Correlation between anti- oxidative stress marker SOD and pain intensity | 7 days
  A negative correlation between concentration of anti-oxidative stress marker SOD and pain intensity (VAS score) in postoperatively in surgically treated patients with laryngeal cancer is expected.
  The concentrations of anti-oxidative stress marker SOD (pg/mL) in the blood serum were determined by ELISA kits, according to the manufacturer's instructions.
  Pain intensity would be assessed using the visual analog scale (VAS). Scores were based on self-reported measures of pain severity recorded with a mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale (0 mm on the left end of the scale marks ''no pain'' and 100mm on the right end of the scale marks ''the worst pain'').
  Correlation would be calculated with Spearman's rank correlation coefficient.
Correlation between anti- oxidative stress marker GPX1 and pain intensity | 7 days
  A negative correlation between concentration of anti- oxidative stress marker GPX1 and pain intensity (VAS score) in postoperatively in surgically treated patients with laryngeal cancer is expected.
  The concentrations of anti-oxidative stress marker GPX1 (pg/mL) in the blood serum were determined by ELISA kits, according to the manufacturer's instructions.
  Pain intensity would be assessed using the visual analog scale (VAS). Scores were based on self-reported measures of pain severity recorded with a mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale (0 mm on the left end of the scale marks ''no pain'' and 100mm on the right end of the scale marks ''the worst pain'').
  Correlation would be calculated with Spearman's rank correlation coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Ana D Jotic, MD, PhD, Study Director — Clinic for otorhinolaryngology and maxillofacial surgery, Clinical center of Serbia; Katarina R Savic Vujovic, MD, PhD, Study Director — Clinical Pharmacology and Toxicology, Faculty of Medicine, University of Belgrade
Locations (2):
- Serbia (2):
  - Clinic for otorhinolaryngology and maxillofacial surgery, Clinical Center of Serbia, Belgrade
  - Clinical Pharmacology and Toxicology, Faculty of Medicine, University of Belgrade, Belgrade

IPD SHARING:
Plan to Share IPD: Yes
Available and ethical compliant patients data will be submitted to the data repository
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months after completion of the study
Access Criteria: Interested investigators can access the data through available link

REFERENCES:
- [Background] Hinther A, Nakoneshny SC, Chandarana SP, Wayne Matthews T, Dort JC. Efficacy of postoperative pain management in head and neck cancer patients. J Otolaryngol Head Neck Surg. 2018 May 2;47(1):29. doi: 10.1186/s40463-018-0274-y. PMID 29720267
- [Background] Sies H, Berndt C, Jones DP. Oxidative Stress. Annu Rev Biochem. 2017 Jun 20;86:715-748. doi: 10.1146/annurev-biochem-061516-045037. Epub 2017 Apr 24. PMID 28441057
- [Background] Niklander SE, Murdoch C, Hunter KD. IL-1/IL-1R Signaling in Head and Neck Cancer. Front Oral Health. 2021 Aug 26;2:722676. doi: 10.3389/froh.2021.722676. eCollection 2021. PMID 35048046
- [Result] Purdy M, Karkkainen J, Kokki M, Anttila M, Aspinen S, Juvonen P, Kokki H, Pulkki K, Rantanen T, Eskelinen M. Does Rectus Sheath Block Analgesia Alter Levels of the Oxidative Stress Biomarker Glutathione Peroxidase: A Randomised Trial of Patients with Cancer and Benign Disease. Anticancer Res. 2017 Feb;37(2):897-902. doi: 10.21873/anticanres.11396. PMID 28179349
- [Result] Salzman R, Kankova K, Pacal L, Tomandl J, Horakova Z, Kostrica R. Increased activity of superoxide dismutase in advanced stages of head and neck squamous cell carcinoma with locoregional metastases. Neoplasma. 2007;54(4):321-5. PMID 17822322
- [Result] Uz U, Eskiizmir G. Association Between Interleukin-6 and Head and Neck Squamous Cell Carcinoma: A Systematic Review. Clin Exp Otorhinolaryngol. 2021 Feb;14(1):50-60. doi: 10.21053/ceo.2019.00906. Epub 2021 Feb 1. PMID 33587847
- [Result] Rettig TC, Verwijmeren L, Dijkstra IM, Boerma D, van de Garde EM, Noordzij PG. Postoperative Interleukin-6 Level and Early Detection of Complications After Elective Major Abdominal Surgery. Ann Surg. 2016 Jun;263(6):1207-12. doi: 10.1097/SLA.0000000000001342. PMID 26135695
- [Result] Karkkainen J, Selander T, Purdy M, Juvonen P, Eskelinen M. Patients with Increased Levels of the Oxidative Stress Biomarker SOD1 Appear to Have Diminished Postoperative Pain After Midline Laparotomy: A Randomised Trial with Special Reference to Postoperative Pain Score (NRS). Anticancer Res. 2018 Feb;38(2):1003-1008. doi: 10.21873/anticanres.12315. PMID 29374733
- [Result] Liu Q, Xu K. Evaluation of some cellular biomarker proteins, oxidative stress and clinical indices as results of laparoscopic appendectomy for perforated appendicitis in children. Cell Mol Biol (Noisy-le-grand). 2020 Jun 5;66(3):197-203. PMID 32538771
- [Result] Si HB, Yang TM, Zeng Y, Zhou ZK, Pei FX, Lu YR, Cheng JQ, Shen B. Correlations between inflammatory cytokines, muscle damage markers and acute postoperative pain following primary total knee arthroplasty. BMC Musculoskelet Disord. 2017 Jun 17;18(1):265. doi: 10.1186/s12891-017-1597-y. PMID 28623906
- [Result] Xi MY, Li SS, Zhang C, Zhang L, Wang T, Yu C. Nalbuphine for Analgesia After Orthognathic Surgery and Its Effect on Postoperative Inflammatory and Oxidative Stress: A Randomized Double-Blind Controlled Trial. J Oral Maxillofac Surg. 2020 Apr;78(4):528-537. doi: 10.1016/j.joms.2019.10.017. Epub 2019 Nov 5. PMID 31785250
- [Result] Liu D, Liu H, Wu J, Gong B. Effects of Thoracic Paravertebral Blockon Inflammatory Response, Stress Response, Hemodynamics and Anesthesia Resuscitation inGallbladder Carcinoma. Cell Mol Biol (Noisy-le-grand). 2022 Feb 28;68(2):171-177. doi: 10.14715/cmb/2022.68.2.24. PMID 35869710
- [Derived] Zivkovic A, Jotic A, Dozic I, Randjelovic S, Cirkovic I, Medic B, Milovanovic J, Trivic A, Korugic A, Vukasinovic I, Savic Vujovic K. Role of Oxidative Stress and Inflammation in Postoperative Complications and Quality of Life After Laryngeal Cancer Surgery. Cells. 2024 Nov 23;13(23):1951. doi: 10.3390/cells13231951. PMID 39682700